CLINICAL TRIAL: NCT05817214
Title: Cadonilimab Plus Anlotinib for Recurrent, Metastasis or Persistent Cervical Cancer
Brief Title: Cadonilimab Plus Anlotinib for R/M/P Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Collaborators: Akeso Biopharma Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Hui Qiu, Chief of Department of Radiation and Medical Gynecologic Oncology, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-01
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cadonilimab; Anlotinib; Granulocyte-macrophage colony-stimulating factor; Immunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — anlotinib; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): This trial has a single treatment arm. All participants will receive small treatment including cadonilimab, anlotinib and granulocyte-macrophage colony-stimulating factor in this arm
  Interventions: Drug: Cadonilimab; Drug: Anlotinib; Drug: Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Drug: Cadonilimab — All Participants will receive cadonilimab of 10mg/kg every three weeks at day 1
  Other Names: AK104
Drug: Anlotinib — All Participants will take anlotinib (12mg) orally in day 1 to day 14, then take a 7 days break.
  Other Names: AL001
Drug: Granulocyte-Macrophage Colony-Stimulating Factor — All Participants will have subcutaneously injection of granulocyte-macrophage colony-stimulating factor from day 1 to day 14, then take a 7 days break.

SUMMARY:
The goal of this clinical trial is to test a new treatment combination including cadonilimab, anlotinib and granulocyte-macrophage colony-stimulating factor (GM-CSF) in recurrent, metastasis and persistent cervical cancer. The main questions it aims to answer are:

* The efficacy of this combination in R/M/P CC;
* The tolerance of this combination in R/M/P CC;
* Possible biomarker of treatment response for this combination.

Participants will receive cadonilimab of 10mg/kg every three weeks at day 1, take anlotinib (12mg) orally in day 1 to day 14, then take a 7 days break and subcutaneously injection of GM-CSF (200ug) from day 1 to day 14, then also take a 7-days break. This treatment will continue until progression or intolerable toxicity or withdraw of participants and it will last for no longer than 2 years.

DETAILED DESCRIPTION:
The prognosis was poor for recurrent, metastasis and persistent cervical cancer especially for those who had multiple lesions and history of previous radiation therapy. KEYNOTE-826 Study demonstrated survival benefit of adding pembrolizumab into the standard first-line treatment for cervical cancer. Here we designed a exploratory clinical study to test a new treatment combination including cadonilimab and anlotinib in recurrent, metastasis and persistent cervical cancer. All participants will receive cadonilimab of 10mg/kg every three weeks at day 1, take anlotinib (8mg) orally in day 1 to day 14, then take a 7-days break and subcutaneously injection of GM-CSF (200ug) from day 1 to day 14, then also take a 7-days break. This treatment will continue until progression or intolerable toxicity or withdraw of participants and it will last for no longer than 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent signed by the patient or their legal representative;
2. Female patients aged ≥18 and ≤75 years old;
3. ECOG PS score of 0-1;
4. Expected survival period ≥6 months;
5. Pathological types include squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma originating from the cervix;
6. Can provide tumor tissue specimens archived within 2 years or willing to undergo tumor tissue biopsy to provide fresh specimens for further testing;
7. At least one evaluable lesion meeting the criteria of RECIST 1.1;
8. Have only received standard first-line systemic treatment in the past: (1) If first-line treatment does not include immunotherapy, failure of first-line treatment is sufficient (for patients who have previously achieved cure, any number of neoadjuvant or adjuvant chemotherapy cycles do not count towards the line count, unless disease progression occurs within 3 months after ≥3 cycles of neoadjuvant/adjuvant chemotherapy; for persistent disease, ≥2 cycles of previous chemotherapy can be counted as one line, otherwise not counted); (2) If first-line treatment includes immunotherapy, clinical benefit must occur after first-line treatment, namely partial or complete tumor remission, with the duration of efficacy lasting more than 6 months.
9. Sitting blood pressure in a resting state is below the normal high value (<140/90 mmHg), or 24-hour dynamic blood pressure monitoring average blood pressure is below the normal high value (<140/90 mmHg), regardless of whether antihypertensive drugs are being taken orally;
10. Hematological indicators meet the following criteria (not transfused or administered hematopoietic growth factor drugs within the past 7 days): white blood cell count (WBC) ≥3.5×109/L, absolute neutrophil count (ANC) ≥1.5×109/L, platelets (PLT) ≥100×109/L, hemoglobin (Hb) ≥90g/L;
11. Liver function indicators meet the following criteria: ALT and AST ≤2.5 times the upper limit of normal (ULN), bilirubin ≤1.5×ULN, albumin ≥35g/L;
12. Coagulation function indicators meet the following criteria (not receiving anticoagulant or hemostatic drug therapy): PT and APTT ≤1.5×ULN, while INR ≤1.5 ULN;
13. Renal function indicators meet the following criteria: blood urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN, urinary protein <2+ or 24-hour urinary protein quantification <1g;
14. Women of childbearing age must undergo serum pregnancy testing within 7 days before initial medication, with negative results, and not be lactating. Female subjects of childbearing age must agree to use effective contraception during the study period and within 180 days after the last dose of the study drug;
15. Good compliance.

Exclusion Criteria:

Translation:

1. Any unstable systemic diseases, including but not limited to active infections within 4 weeks (defined as fever exceeding 38.5°C, evidence of bacteremia, or evidence of infectious changes in the heart, brain, kidneys, lungs, liver, and intestines), circulatory accidents within 6 months (malignant hypertensive crisis, myocardial infarction, severe/unstable angina, heart failure above NYHA class 2, clinically significant supraventricular or ventricular arrhythmias, or cerebral vascular accidents not yet recovered from or resulting in severe sequelae), uncontrolled type 2 diabetes (fasting blood glucose >11.1 mmol/L or glycated hemoglobin >8%), and pulmonary insufficiency (any cause leading to decreased lung function, defined as FEV1/FVC <70%, FEV1 <80% of predicted value).
2. History of autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, autoimmune liver diseases, systemic vasculitis, scleroderma, dermatomyositis, autoimmune hemolytic anemia;
3. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; hepatitis C, defined as HCV-RNA higher than the detection limit of the assay) or combined hepatitis B and hepatitis C infection;
4. History of attenuated live vaccine administration within 28 days before the first dose of the study drug or expected attenuated live vaccine administration during the study period;
5. Tumor invasion of major blood vessels on imaging or investigator judgment indicating a high risk of tumor invasion of important vessels causing fatal bleeding or other diseases with a high risk of severe bleeding;
6. Previous treatment with anlotinib or cadonilimab;
7. Evidence of active tuberculosis infection within the past year before screening;
8. Diagnosis of any other malignant tumors, adequately treated basal cell carcinoma or squamous cell skin carcinoma, or cervical carcinoma in situ within 5 years before entering the study;
9. Major surgery within 28 days before randomization (tissue biopsy for diagnostic purposes and insertion of a central venous catheter via percutaneous puncture are allowed);
10. Active venous or arterial thromboembolic events within 6 months before randomization, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism;
11. Previous or planned allogeneic bone marrow or solid organ transplantation;
12. Clinically significant intestinal obstruction, occurrence of intestinal repair, intestinal anastomosis, intestinal diversion, or enterocutaneous fistula for any reason at any time;
13. Participants who experienced symptoms of hemoptysis within 2 months before entering the study and had a maximum daily hemoptysis volume of approximately ≥2.5 mL. Participants who experienced significant bleeding symptoms or had a clear bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcers, baseline fecal occult blood test ++ and above, or vasculitis, within 3 months before entering the study; known hereditary or acquired bleeding and thrombotic tendencies, such as hemophilia, coagulation disorders, thrombocytopenia, splenic hyperfunction, etc.;
14. Visible hematuria or other evidence of active urinary system bleeding;
15. Currently receiving thrombolysis or requiring long-term anticoagulant therapy with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day);
16. Known allergy to anlotinib, cadonilimab or any of their excipients;
17. Participation in any other drug clinical studies within the previous 4 weeks before randomization or within 5 half-lives of the last study drug administration;
18. History of substance abuse, alcoholism, or drug addiction;
19. Coexisting severe cognitive impairment and inability to achieve stable mental status;
20. As judged by the investigator, patients may have other factors that could lead to premature termination of the study, such as other serious illnesses or severe laboratory abnormalities, or factors affecting the safety of the participants or the collection of trial data and samples due to family or social reasons, etc.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 2 years
  Rate of participants with complete response plus partial response as best response in the intent to treatment group according to RECIST 1.1

SECONDARY OUTCOMES:
Rate and grade of adverse events | From enrollment to 90 days after last treatment of all subjects
  The incidence of adverse events and severity graded according to CTCAE 5.0
Disease control rate | up to 2 years
  Rate of participants with complete response plus partial response plus stable disease as best response in the intent to treatment group according to RECIST 1.1
Duration of Response | Up to 2 years
  Time period from first response to first progression
Progression free survival rate | Up to 2 years
  Proportion of participants without tumor recurrence or death
Overall survival rate | Up to 2 years
  Proportion of survival participants

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qiu, Ph.D., Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No